CLINICAL TRIAL: NCT05055167
Title: A Phase II Study of Envafolimab as First-line Treatment of Aged Patients With High PD-L1 Expression Stage in Advanced Non-small-cell Lung Cancer(NSCLC)
Brief Title: Envafolimab as First-line Treatment of Aged Patients in Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-006
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab (Experimental): Elderly NSCLC Patients with high PD-L1 expression
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab — single agent, 300mg Q3W IH until disease progressed

SUMMARY:
Explore the efficacy and safety of Envafolimab in first line treatment of elderly patients with locally advanced or metastatic non-small cell lung cancer with high PD-L1 expression, view to providing better treatment options for elderly patients with high PD-L1 expression and improving the survival and prognosis of patients .

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age strictly at least 70 years.
* Cytologically or histologically proven NSCLC(adenocarcinoma, epidermoid carcinoma, large-cell carcinoma) of locally advanced (stage IIIb/IIIc), metastatic, or relapsing (stage IV) according to the American Joint Committee on Cancer Staging Handbook.
* Presence of at least one measurable target lesion (RECIST rules) in a non irradiated region.
* No previous systemic chemotherapy for lung cancer.
* PD-L1≥50% in tissue samples detected by immunohistochemistry.
* PS 0 or 1.
* Life expectancy sup 12 weeks.
* Normal hematologic function.

Exclusion Criteria:

* EGFR-sensitive mutations or ALK rearrangements
* Previous treatment with immune checkpoint inhibitors
* Presence of symptomatic brain metastases；
* Chinese patent medicine with anti-lung cancer indications or immunoregulatory drugs (including thymopeptide, interferon and interleukin, except for the local use of pleural effusion control) for systemic treatment；
* Another previous or concomitant cancer, except for basocellular cancer of the skin or treated cervical cancer in situ；
* Concurrent administration of one or several other antitumor therapies；
* Concurrent participation in another clinical trial；
* Active autoimmune disease requiring systemic treatment occurred within 2 years prior to initial；
* Systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to initial administration；
* Contraindication to the study drugs；
* Has not fully recovered from toxicity and/or complications caused by any intervention prior to the commencement of treatment (i.e., grade 1 or baseline, excluding fatigue or hair loss);
* A history of human immunodeficiency virus (HIV) infection;
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the research center);
* Active HCV infected;
* Recent vaccination within 30 days before the first administration (cycle 1, day 1);
* Other severe concurrent disorders that occurred during the prior six months before enrollment (myocardial infection, severe or unstable angor, NYHA class 3 or 4 congestive heart failure, transient or constituted cerebral ischemic attack, psychiatric or neurological disorders preventing the patient from understanding the trial, uncontrolled infections).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 48 months
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of Almonertinib to the end of study.

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No